CLINICAL TRIAL: NCT00171262
Title: Trial to Evaluate the Efficacy of Fluvastatin on Certain Markers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CXUO320BES02
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Dyslipidemia
Keywords: Dyslipidemia, chronic renal disease, fluvastatin
MeSH Terms: conditions — Dyslipidemias; Renal Insufficiency, Chronic | interventions — Fluvastatin

INTERVENTIONS:
Drug: Fluvastatin

SUMMARY:
To analyze efficacy of fluvastatin on patients with chronic renal disease by analyzing certain inflammatory markers. In addition, tolerability and safety will also be evaluated in a Spanish population.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years Patients that give their inform consent

Exclusion Criteria:

* Pregnant women Diabetic patients Treated with statins for the year prior to study inclusion Patients with contraindications listed in fluvastatin prescribing information

Other protocol-defined in and exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in serum inflammatory markers after 52 weeks

SECONDARY OUTCOMES:
Change from baseline in fibrosis parameters and endothelial function after 52 weeks
Adverse events and serious adverse events after 52 weeks
Change from baseline in laboratory tests of kidney function after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Madrid, Spain